CLINICAL TRIAL: NCT01336062
Title: Phase Ib/IIa, Two-stage Trial of ABI-007 Plus S-1 as Second-line Chemotherapy in Advanced Gastric Cancer Patients
Brief Title: Trial of ABI-007 Plus S-1 as Second-line Chemotherapy in Advanced Gastric Cancer Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, PRO., Peking University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NAB-PTX-GC
Record Dates: First submitted 2011-04-04; First posted 2011-04-15 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Gastric Adenocarcinoma
Keywords: advanced; resistant to prior chemotherapy
MeSH Terms: interventions — Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nanoparticle Albumin-Bound Paclitaxel (Experimental): The study evaluate 3 dose level of nab-paclitaxel:100 mg /m2;125 mg /m2;80 mg /m2;
  Interventions: Drug: Nanoparticle Albumin-Bound Paclitaxel

INTERVENTIONS:
Drug: Nanoparticle Albumin-Bound Paclitaxel — this study evaluate 3 dose level of nab-paclitaxel:100 mg /m2;125 mg /m2;80 mg /m2;

SUMMARY:
Gastric cancer have poor prognosis and majority of patients resistant to 5-FU/DDP based first-line chemotherapy in China. There was no recommended second-line chemotherapy for advanced gastric cancer. Taxane is promising in gastric cancer. Nanoparticle Albumin-Bound Paclitaxel (Abraxane，ABI-007) has good convenience to use and been approved in breast cancer in many countries. The investigator then initiated a prospective phase Ib/IIa clinical trial with nab-paclitaxel plus TS-1 as the second-line treatment in advanced gastric cancer to observe the safety and efficacy.

DETAILED DESCRIPTION:
This study is a two-stage design. Stage 1

The investigator should evaluate two recommend dose and tolerability of nab-paclitaxel plus S-1 after one course of treatment as 3+1 design:

nab-paclitaxel should be given intravenously on days 1 and 8 at a dose as follows, Treatment should be repeated every 3 weeks: Treatment arm A：125 mg /m2; Treatment arm B：100 mg /m2; Treatment arm C: 80 mg /m2; S-1 should be given orally twice a day as follows for 14 consecutive days, followed by a 1-week rest. Treatment should be repeated every 3 weeks. BSA < 1.5 m2，40mg，bid;BSA ≥ 1.5 m2，50mg，bid.

The investigator should determine whether to continue the original regimen; compare the safety and pharmacokinetic results with original profile of combination therapy to select the best therapy programs (RD, recommended dose).

Stage 2 According to two-stage design (Simon,1989), re-entry subjects to the recommended dose group to a total of 25 valid cases. If 11 patients achieve response, then enter the second phase of total 66 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form
2. Age 18-75 years;
3. Histologically or cytologically confirmed gastric cancer;
4. Advanced or recurrent, metastatic disease;
5. Performance Status- Eastern Cooperative Oncology Group (ECOG) 0-1;
6. Life expectancy of at least 12 weeks;
7. At least have one measurable disease(according to RECIST, Response Evaluation Criteria in Solid Tumors )
8. Subjects who have received one prior regimen for gastric carcinoma and developed disease progression or recurrence within 6 months after the end of systemic adjuvant treatment. The regimen must have contained fluorouracil(e.g. 5-FU,capecitabine) and/or cisplatin;
9. Haematopoietic status:

   * Absolute neutrophil count > 1.5 x 109/L,
   * Platelet count > 90 x 109/L,
   * Hemoglobin at least 9 g/dl,
10. Hepatic status:

    * Bilirubin ≤ 1.5 x upper limit of normal (ULN),
    * AST and ALT ≤ 2.5 times ULN(no liver metastasis), ≤5 times ULN(with liver metastasis)
11. Renal status:

    - Creatinine ≤1.5 times ULN or calculated creatinine clearance, using the Cockcroft-Gault formula, ≥40 mL/min;
12. Able to swallow and retain oral medication；without malabsorption syndrome, or disease significantly affecting gastrointestinal function, such as ulcerative colitis and Crohn's disease;
13. Cardiovascular: Baseline LVEF 50% measured by echocardiography (ECHO) ;
14. Negative serum pregnancy test (For women of childbearing potential);Fertile patients must use effective contraception.

Exclusion Criteria:

1. Received any prior treatment including taxane or S-1;
2. Concurrent systemic anti-cancer therapy (immunotherapy, biologic therapy, hormone therapy, etc ); received treatment with an investigational agent or participation in another therapeutic clinical trial within 4 weeks;
3. Unresolved or unstable, serious toxicity from prior cancer treatment (any toxicities greater than grade 2; peripheral neuropathy of grade 2 or greater
4. Symptomatic brain metastasis;
5. Known history of uncontrolled or symptomatic angina, clinically significant arrhythmias, congestive heart failure, uncontrolled hypertension (≥ 180/110), unstable diabetes mellitus, dyspnea at rest, or chronic therapy with oxygen;
6. History of other malignancy. However, subjects with a past or current history of completely resected basal and squamous cell carcinoma of the skin or successfully treated in situ carcinoma of the cervix are eligible
7. Dementia, altered mental status, or any psychiatric condition that would prevent the understanding or rendering of ICF;
8. Active or uncontrolled infection;
9. Concurrent treatment with an investigational agent or participation in another therapeutic clinical trial;
10. Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
adverse events | during the treatment in the hosptital,an expected average of 3 weeks
  participants will be followed for the duration of hospital stay, an expected average of 3 weeks
Objective response rate | 6 weeks
  CT/MRI will be performed every 2 cycles of treatment for efficacy evaluation

SECONDARY OUTCOMES:
progression free survival | 1 year
  the follow-up visit of PFS will be performed every 6 weeks
overall survival of participants | 2 years
  OS means that from the first dose of treatment drug to death or lost, the follow-up visit will be performed every 3 months till death or lost
biomarkers | 6 weeks
  If the tumour samples available, to identify the molecular characteristics(such as SPARK,ABCG2,β-Tubulin III,PDGFRA,etc) of responding tumours by immunohistochemical, FISH, genomic and proteomic analysis; To study biomarkers expression before and during therapy and establish correlations with clinical outcome and toxicity;

CONTACTS AND LOCATIONS:
Locations (1):
- Lin Shen, Beijing, Beijing Municipality, China